CLINICAL TRIAL: NCT02028000
Title: Post-Operative Pain and Skin Closure Methods After Cesarean Section
Brief Title: Postoperative Pain and Skin Closure Methods After Cesarean Section
Acronym: Skin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient data to continue. Study will not resume.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17928
Record Dates: First submitted 2012-10-09; First posted 2014-01-06 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Pregnancy
Keywords: Pregnancy; Pregnant; Cesarean Section Delivery

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- INSORB staples skin closure (Active Comparator): Women undergoing cesarean section delivery will have skin closure with INSORB staples.
  Interventions: Procedure: Monocryl skin closure; Procedure: Vicryl skin closure
- Monocryl skin closure (Active Comparator): Women undergoing cesarean section delivery will have skin closure with Monocryl.
  Interventions: Procedure: Insorb staples skin closure; Procedure: Vicryl skin closure
- Vicryl skin closure (Active Comparator): Women undergoing cesarean section delivery will have Vicryl skin closure
  Interventions: Procedure: Insorb staples skin closure; Procedure: Monocryl skin closure

INTERVENTIONS:
Procedure: Insorb staples skin closure — Patients will be randomized to Insorb staples skin closure and compared to Monocryl and Vicryl group.
  Arms: Monocryl skin closure; Vicryl skin closure
Procedure: Monocryl skin closure — Patients will be randomized to Monocryl skin closure and compared to Insorb skin closure and Vicryl skin closure.
  Arms: INSORB staples skin closure; Vicryl skin closure
Procedure: Vicryl skin closure — Patients will be randomized to Vicryl skin closure and compared to Insorb and Monocryl skin closure groups.
  Arms: INSORB staples skin closure; Monocryl skin closure

SUMMARY:
The study is looking at women undergoing cesarean section delivery of their baby. The purpose of this research study is to determine what type of skin closure after cesarean section helps decrease pain level the most and improves the appearance of the incision site.

The study hypothesis is to determine if skin closure with absorbable subcuticular staples leads to improved cosmesis and/or decreased post-operative pain.

Participants in the study will already be scheduled for a cesarean section for delivery of their baby. They will be randomized into one of three groups, 1) Insorb (absorbable subcuticular stapes), 2) Vicryl suture or 3) Monocryl suture for the skin closure of their cesarean section. Information that will be recorded includes amount of pain medication usage while in the hospital after cesarean section, daily patient rated pain score until discharge from hospital, pain score 6 weeks after surgery and cesarean section cosmetic scar 6 weeks after surgery.

DETAILED DESCRIPTION:
Cesarean delivery is the most common surgical procedure performed in the United States, with over 1 million procedures performed per year. Based on recent Centers for Disease Control National Vital Statistics Report 32.3% of all births in the United States were via cesarean delivery, marking the twelfth consecutive annual increase in the cesarean delivery rate. Given the high numbers of cesarean deliveries being performed today, there has been interest in optimizing surgical techniques. Several recent reviews have summarized the evidence for various steps of cesarean delivery, but surprisingly in many cases there is little scientific evidence on which to base the choice of surgical technique.

The topic of skin closure after cesarean delivery is an area that has been the focus of several randomized control trials. The trials compared surgical steel staples to subcuticular suture of various materials focusing on differences in post-operative pain, infection rates, and scar cosmesis. Cosmesis has been investigated in all three Randomized Clinical Trials and none have found differences between surgical steel staples and subcuticular suture. Infection rate has been studied in a single observational study which found a higher infection rate in those patients whose skin was closed with surgical steel staples compared to suture. Studies of post-operative pain and skin closure technique have been contradictory. The earliest Randomized clinical trial to investigate skin closure and post-operative pain was done by Frishman et al (5) and found that subjective self-assessment of pain was better at hospital discharge and 6 weeks post-operatively in patients when subcuticular suture rather than surgical steel staples were used. A subsequent Randomized clinical trial reported the opposite result with less pain 6 weeks post-operatively when surgical steel staples were used. This discrepancy may, in part, be due to the different suture material used in the two trials. The study by Frishman et al which showed a benefit of subcuticular suture utilized used polyglycolic acid (Vicryl suture or Insorb staples); whereas, the study by Rousseau et al used polyglecaprone (Monocryl suture). To date direct comparison of skin closure at the time of cesarean with these two suture materials has not been performed.

Recently, a new technology for skin closure has been introduced that employs absorbable material, polylactic and polyglycolic acid, in subcuticular staples. In animal models this method of skin closure has shown less histological inflammation and fewer wound infections than either surgical steel staples or subcuticular suture. Unfortunately, little is known about how this skin closure technique compares to the other more established techniques after cesarean delivery in humans. However, a retrospective analysis comparing subcuticular absorbable staples with surgical steel staples revealed an association between subcuticular absorbable staples and decreased in-hospital analgesic use. The current study is a prospective randomized trial that investigates four cesarean skin closure techniques-surgical steel staples, subcuticular polyglycolic acid suture (Vicryl), subcuticular, polyglecaprone suture (Monocryl), and absorbable subcuticular polyglycolic acid staples-to determine if one is associated with improved cosmesis or a decrease in post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-44
* Any race
* Any parity
* Scheduled Cesarean Section
* Neuraxial analgesia

Exclusion Criteria:

* Diabetes Mellitus
* Maternal Connective Tissue Disorder
* Maternal Steroid Use

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
Intravenous and analgesic use. | Admission for delivery of baby by cesarean section to expected postpartum average of 6 weeks
  Record the amount of in hospital intravenous and oral analgesic use.
Daily subjective pain score while hospitalized | Hospital admission for cesarean section delivery
  Daily patient rated subjective pain score (0-10 based on visual analog scale) until dismissal from the hospital will be recorded.
6 week postoperative subjective pain score | After cesarean section delivery at the 6 week postpartum visit
  Patient rated subjective pain score 6 weeks postoperatively will be recorded.
Scar cosmetic score 6 weeks post-operatively. | 6 weeks post-operatively after cesarean section
  6 weeks post-operative scar cosmetic score will be recorded.

SECONDARY OUTCOMES:
Wound complications | Time of cesarean section until 6 weeks postpartum visit
  Wound complications (infection, separation, or seroma)
Length of hospital stay | C/S admission to discharge time
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Nitsche, MD, PhD, Principal Investigator — Wake Forest Baptist School of Medicine
Locations (1):
- Forsyth Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Walsh CA. Evidence-based cesarean technique. Curr Opin Obstet Gynecol. 2010 Apr;22(2):110-5. doi: 10.1097/GCO.0b013e3283372327. PMID 20216417
- [Background] Johnson A, Young D, Reilly J. Caesarean section surgical site infection surveillance. J Hosp Infect. 2006 Sep;64(1):30-5. doi: 10.1016/j.jhin.2006.03.020. Epub 2006 Jul 5. PMID 16822582
- [Background] Pineros-Fernandez A, Salopek LS, Rodeheaver PF, Drake DB, Edlich RF, Rodeheaver GT. A revolutionary advance in skin closure compared to current methods. J Long Term Eff Med Implants. 2006;16(1):19-27. doi: 10.1615/jlongtermeffmedimplants.v16.i1.30. PMID 16566742
- [Background] Hamilton BE, Martin JA, Ventura SJ. Births: preliminary data for 2009. Natl Vital Stat Rep. 2010 Dec;59(3):1-19. PMID 25073731
- [Result] Altman AD, Allen VM, McNeil SA, Dempster J. Pfannenstiel incision closure: a review of current skin closure techniques. J Obstet Gynaecol Can. 2009 Jun;31(6):514-520. doi: 10.1016/S1701-2163(16)34213-X. PMID 19646316
- [Result] Berghella V, Baxter JK, Chauhan SP. Evidence-based surgery for cesarean delivery. Am J Obstet Gynecol. 2005 Nov;193(5):1607-17. doi: 10.1016/j.ajog.2005.03.063. PMID 16260200
- [Result] Frishman GN, Schwartz T, Hogan JW. Closure of Pfannenstiel skin incisions. Staples vs. subcuticular suture. J Reprod Med. 1997 Oct;42(10):627-30. PMID 9350017
- [Result] Gaertner I, Burkhardt T, Beinder E. Scar appearance of different skin and subcutaneous tissue closure techniques in caesarean section: a randomized study. Eur J Obstet Gynecol Reprod Biol. 2008 May;138(1):29-33. doi: 10.1016/j.ejogrb.2007.07.003. Epub 2007 Sep 6. PMID 17825472
- [Result] Rousseau JA, Girard K, Turcot-Lemay L, Thomas N. A randomized study comparing skin closure in cesarean sections: staples vs subcuticular sutures. Am J Obstet Gynecol. 2009 Mar;200(3):265.e1-4. doi: 10.1016/j.ajog.2009.01.019. PMID 19254586
- [Result] Fick JL, Novo RE, Kirchhof N. Comparison of gross and histologic tissue responses of skin incisions closed by use of absorbable subcuticular staples, cutaneous metal staples, and polyglactin 910 suture in pigs. Am J Vet Res. 2005 Nov;66(11):1975-84. doi: 10.2460/ajvr.2005.66.1975. PMID 16334959
- [Result] Singer AJ, Arora B, Dagum A, Valentine S, Hollander JE. Development and validation of a novel scar evaluation scale. Plast Reconstr Surg. 2007 Dec;120(7):1892-1897. doi: 10.1097/01.prs.0000287275.15511.10. PMID 18090752